CLINICAL TRIAL: NCT02103855
Title: Calcineurin Inhibitors to Belatacept Switch Study to Prevent the Progression of Kidney Disease in Pancreas Transplant Alone Recipients
Brief Title: Switch From Calcineurin Inhibitor to Belatacept in Pancreas Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Asif Sharfuddin, Asif A Sharfuddin, MD, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMS 103-337
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Nephrotoxicity
Keywords: pancreas transplantation; immunosuppression; belatacept
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- belatacept (Experimental): Belatacept 5 mg/kg IVPB q 2 wks x 5 doses followed by 5 mg/kg IVPB q month. The belatacept dose will be infused IV over 30 minutes.
  Day 14: Reduce tacrolimus dose by 25% Day 30: Reduce tacrolimus dose by additional 25% Day 45: Reduce tacrolimus dose by additional 25% Day 60: Stop tacrolimus.
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept
  Other Names: Nulojix

SUMMARY:
Kidney damage is a major complication of current antirejection medicines used in transplantation. An increasing number of brittle diabetics are successfully receiving a pancreas transplant. One of the challenges following pancreas transplant is that a patient can develop kidney damage from one of their antirejection medicines, tacrolimus. The objective of this study is to substitute a new antirejection medicine which does not cause kidney damage, belatacept for tacrolimus in patients that have developed signs of tacrolimus related kidney damage to slow the progression of kidney disease.

DETAILED DESCRIPTION:
Nephrotoxicity is a major complication of current immunosuppression regimens used in transplantation. Pancreas transplantation has been increasedly performed to manage labile diabetes mellitus during the last few decades and survival rates of pancreatic grafts are improving. One of the challenges that is faced following pancreas transplantation alone are pathologic changes from diabetes frequently seen in native kidneys in the pancreas transplant recipients. High levels of calcineurin inhibitors (CNI) have been identified as risk factors for decline in kidney function and progression to end-stage renal disease. The objective of this trial is to take subjects who have biopsy proven CNI toxicity off of their CNI and begin belatacept, which is not a CNI.

The hypothesis is by switching the pancreas transplant subject with documented CNI kidney toxicity to belatacept will slow the progression of chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Pancreas transplant alone recipients
* EBV IgG positive
* Biopsy proven calcineurin inhibitor toxicity on native kidney biopsy
* Maintained on a regimen of tacrolimus, sirolimus, mycophenolate

Exclusion Criteria:

* EBV IgG negative
* Not maintained on an immunosuppression regimen that contains tacrolimus
* Unable or unwilling to give informed consent
* Active infection
* History of malignancy post transplant
* Glomerular filtration rate < 15 mL/min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asif Sharfuddin, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Health, University Hospital, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled and started on June 3, 2014. Last patient enrolled and started on Aug 6, 2014.
  All patients enrolled at Indiana University Hospital - Transplant Unit.
Pre-assignment Details: Participants were enrolled according to inclusion and exclusion criteria. Tacrolimus was weaned according to protocol.
Groups:
- Belatacept: Belatacept 5 mg/kg IVPB q 2 wks x 5 doses followed by 5 mg/kg IVPB q month. The belatacept dose will be infused IV over 30 minutes.
  Day 14: Reduce tacrolimus dose by 25% Day 30: Reduce tacrolimus dose by additional 25% Day 45: Reduce tacrolimus dose by additional 25% Day 60: Stop tacrolimus.
  Belatacept
Period: Overall Study
Arm/Group | Belatacept
Started | 6
Completed | 4
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Belatacept
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Estimated Glomerular Filtration Rate (eGFR)
Description: Change in serum eGFR from baseline to 1 year following conversion from tacrolimus to belatacept
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Belatacept
Number analyzed (Participants) | 4
ml/min/1.73m2 | 2.25 (3.35)

2. Primary Outcome: Serum Creatinine at Year 1
Description: Serum Creatinine measured at 1 year after conversion from Tacrolimus to Belatacept.
Time Frame: 1 year
Population: 4 subjects who completed 1 year of Belatacept were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Belatacept
Number analyzed (Participants) | 4
mg/dl | 1.8 (0.2)

3. Secondary Outcome: Number of Participants With Pancreas Transplant Rejection
Description: Pancreas Rejection as measured by serum amylase, serum lipase.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept
Number analyzed (Participants) | 4
Participants | 2

4. Secondary Outcome: Change From Baseline Serum Hemoglobin A1c
Description: Pancreas Transplant Function was measured by assessing change in Pre HbA1c to Post HbA1c at1 year after conversion.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Belatacept
Number analyzed (Participants) | 6
percentage of glycosylated hemoglobin | 5.9 (0.15)

5. Secondary Outcome: Pancreas Transplant Function as Measured by Fasting Serum Glucose Level.
Description: Fasting Serum Glucose level measured at 1 year after conversion from Tacrolimus to Belatacept.
Time Frame: 1 Year
Population: 4 subjects who completed 1 year of Belatacept.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Belatacept
Number analyzed (Participants) | 4
mg/dl | 96.9 (6.3)

ADVERSE EVENTS:
Arm/Group | Belatacept
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1) — Need for Blood Transfusion
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept (N=6)
Nausea (Gastrointestinal disorders) | 5 (5)
Hypertension (Cardiac disorders) | 2 (2) — Uncontrolled HTN
Hyperlipidemia (Endocrine disorders) | 1 (1)
Hot Flash (Endocrine disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3) — Not needing Blood transfusion
Infection (Infections and infestations) | 3 (3)
Hypokalemia (Renal and urinary disorders) | 1 (1)
Skin Sores (Skin and subcutaneous tissue disorders) | 1 (1)
Retinal Vessel Rupture (Eye disorders) | 1 (1)
Dehydration (Renal and urinary disorders) | 1 (2)
Hair Loss (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No